CLINICAL TRIAL: NCT02027324
Title: Chlorhexidine-Alcohol Vs. Povidone-Iodine for Prevention of Surgical Site Infection After Cesarean Delivery: A Randomized Trial
Brief Title: Prevention of Surgical Site Infection After Cesarean Delivery
Acronym: CAPISSI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Another study with similar methods was recently published
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Arvind Palanisamy, MD, FRCA, Assistant Professor of Anaesthesia, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2013P002037
Record Dates: First submitted 2014-01-02; First posted 2014-01-06 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Surgical Site Infection
Keywords: Surgical site infection; Cesarean delivery; Antisepsis; Povidone iodine; Chlorhexidine alcohol; Endometritis
MeSH Terms: conditions — Surgical Wound Infection; Endometritis | interventions — Chlorhexidine; Ethanol; Population Groups; Povidone-Iodine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chlorhexidine-alcohol group (Experimental): 2% chlorhexidine in 70% isopropyl alcohol in accordance with manufacturer's instructions for safe usage.
  Interventions: Drug: Chlorhexidine-alcohol group
- Povidone-Iodine group (Experimental): 10% Povidone-iodine applied topically according to manufacturer's instructions
  Interventions: Drug: Povidone-Iodine Group

INTERVENTIONS:
Drug: Chlorhexidine-alcohol group — 2% chlorhexidine in 70% isopropyl alcohol in accordance with manufacturer's instructions for safe usage.
  Other Names: Chloraprep
  Arms: Chlorhexidine-alcohol group
Drug: Povidone-Iodine Group — 10% Povidone-Iodine for surgical antisepsis according to manufacturer's instructions.
  Other Names: Betadine
  Arms: Povidone-Iodine group

SUMMARY:
There are approximately 1.4 million cesarean deliveries in the United States each year, and an average of 1250 elective cesarean deliveries each year at the Brigham and Women's Hospital (BWH) in Boston, Massachusetts. Among cesarean deliveries performed at BWH, approximately 2% of patients are diagnosed with a surgical site infection (SSI). Because SSI is associated with significant morbidity and increased cost of care, numerous guidelines exist to guide preoperative administration of prophylactic antibiotics. However, there are no recommendations for the choice of antiseptic solution for prevention of SSI. Among the currently popular antisepsis preparations, chlorhexidine-alcohol (CA) is known to decrease SSI in non-obstetric surgeries. However, the time required for CA to dry (~ 3 min) to minimize flammability risk is disadvantageous in the setting of emergent cesarean delivery. Many institutions use povidone-iodine, another antisepsis preparation that does not require the mandatory drying time. Our randomized study aims to compare the incidence of SSI in patients receiving either CA or PI during elective cesarean delivery, and we hypothesize that CA would be associated with a lower incidence of SSI.

DETAILED DESCRIPTION:
This study will be conducted over three years with an estimated sample size of 4500 patients. Prior to enrollment of study subjects, each year will be divided into 3-month blocks and each block will be assigned one of the two study antiseptic solutions - 2% chlorhexidine gluconate in 70% isopropyl alcohol (CA) or 10% Povidone-Iodine (PI) - in an alternating manner. All patients undergoing elective cesarean deliveries during a block will receive the same preoperative skin preparation, in concordance with guidelines for its use. The block assignments will alternate within each year and the order will be reversed after one year to minimize or eliminate seasonal variation in skin infection rates. All patients will receive routine history and physical examination, blood tests, pre-procedure bathing instructions, and preoperative body hair clipping as desired by their primary obstetric provider. Age, body mass index (BMI), gestational age, history of smoking, previous abdominal surgery, number of pregnancies, and live births will be documented before entry into the study. Eligible patients will receive antibiotic prophylaxis with weight-based cefazolin within 60 min before skin incision. We will collect data on preoperative preparation of the surgical site (clipping vs. shaving), type of skin and uterine incision, method of fascia and skin closure, duration of the procedure, use of postoperative antibiotics, and adverse reactions to the skin preparation. The primary endpoint for this study will be any SSI diagnosed within 30 days of cesarean delivery. Our secondary outcomes will be the type of SSI (based on the Center for Disease Control infection classification) and the time to diagnosis of SSI.

The Infectious Disease department at BWH will perform the surveillance for SSI/endometritis. This team will be blinded to the choice of anti-sepsis preparation during the study period. Briefly, surveillance will include daily, weekly, monthly, and quarterly reviews of data. The infectious disease team will perform a daily review of microbiology results for positive wound and blood cultures, and assess whether the patient had cesarean section within 30 days prior to cultures. On a weekly basis, a report of obstetric patients readmitted within 30 days will be generated, and patients will be selected with an admitting diagnosis consistent with infection in the setting of a history of recent cesarean delivery. Each month, a report of patients will be generated with ICD-9 discharge code for cesarean section as well as ICD-9 codes for other complications of obstetrical surgical wound and major puerperal infection. Post-cesarean delivery patients receiving antibiotics for at least 2 days after the first postoperative day, and those that receive antibiotics during readmission will also be identified and recorded. During every quarter, the number of elective cesarean deliveries performed will be quantified, and the incidence of specific sub-types of SSI (superficial, deep, organ space/endometritis) will be documented. In addition to inpatient surveillance, the electronic clinic records for all patients will be reviewed, and data will be recorded for any SSI that is diagnosed and treated on an outpatient basis. Documentation from discharge to the six-week postpartum visit will be reviewed to ensure data fidelity, but only infections that occur within 30 days of cesarean delivery will be included in the final analyses. Active SSI will be treated according to prevailing guidelines.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for elective cesarean delivery

Exclusion Criteria:

* Allergy to either of the antiseptic preparations
* Ongoing active skin or systemic infection
* Pre-operative antibiotic therapy for non-surgical reasons
* Those unable to receive antibiotic prophylaxis

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of Surgical Site Infection within 30 days of Cesarean Delivery | At 3 years after first patient enrollment

SECONDARY OUTCOMES:
Type of SSI (based on CDC classification) | 3 years after initial enrollment
Time to diagnosis of SSI | 3 years after initial enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Arvind Palanisamy, MD, FRCA, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States